CLINICAL TRIAL: NCT04642261
Title: Effect of Empagliflozin on Liver Fat in Non-alcoholic Fatty Liver Disease Patients Without Diabetes Mellitus: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Empagliflozin on Liver Fat in Non-diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Cheung Ka Shing, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 20-065
Record Dates: First submitted 2020-11-06; First posted 2020-11-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; fatty liver; empagliflozin; SGLT2 inhibitors
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomly allocated to either the empagliflozin group or placebo group (i.e. control group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo pills will be manufactured in identical appearance to the study drug (empagliflozin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin group (Experimental): Empagliflozin 10mg daily for 52 weeks
  Interventions: Drug: Empagliflozin 10 MG
- Placebo group (Placebo Comparator): Placebo pills (identical in appearance to empagliflozin 10mg) daily for 52 weeks
  Interventions: Drug: Placebo pills

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10mg daily
  Other Names: empagliflozin
  Arms: Empagliflozin group
Drug: Placebo pills — Identical in appearance to empagliflozin 10mg daily
  Arms: Placebo group

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a global epidemic with a prevalence of 25%. Currently therapies for NAFLD patients without diabetes mellitus (DM) are limited, and are associated with various adverse side effects. Sodium-glucose cotransporter type-2 (SGLT2) inhibitors can reduce hepatic fat content in patients with DM. However, the role of SGLT2 inhibitors in NAFLD patients without DM has not been investigated. Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) and liver stiffness measurement (LSM) are non-invasive methods to diagnose hepatic steatosis and fibrosis/cirrhosis, respectively.

The investigators propose a double-blind, randomized, placebo-controlled trial to compare the effects of empagliflozin (a type of SLGT2 inhibitors) versus placebo (in a 1:1 ratio) in reducing hepatic fat content as measured by MRI-PDFF in NAFLD patients without DM. A total of 98 adult patients will be randomly sampled from the liver clinic in our local hospital. Empagliflozin 10mg daily will be given to the treatment arm. The placebo pill will be manufactured to be identical in appearance to the study drug. Eligible subjects will be followed up until week 52, and will undergo clinical, anthropometric and laboratory assessments (including liver function test and fasting blood) at baseline, week 6, 12, 26, 40 and 52. They will undergo LSM at baseline, week 26 and 52, and MRI-PDFF at baseline and week 52. The primary outcome will be a difference in change of liver fat content (measured by MRI-PDFF) at week 52 from baseline between the two groups.

The study results will determine whether SGLT2 inhibitors can reduce hepatic steatosis in NAFLD patients without DM.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a global epidemic with a prevalence of 25%. Currently therapies for NAFLD patients without diabetes mellitus (DM) are limited, and are associated with various adverse side effects. Sodium-glucose cotransporter type-2 (SGLT2) inhibitors are antidiabetic drugs that reduce hepatic fat content in patients with DM, which is independent of glycemic control. However, the role of SGLT2 inhibitors in NAFLD patients without DM has not been investigated. Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) is an emerging non-invasive imaging technique, and is more sensitive than liver biopsy/histology in quantifying liver fat change. Liver stiffness measurement (LSM) by transient elastography is a non-invasive method to diagnose fibrosis/cirrhosis with high accuracy.

The novelty of utilizing the concept of "drug repositioning" by changing the role of SGLT2 inhibitors in treating DM to treating NAFLD in patients without DM deserves exploration. The investigators propose a double-blind, randomized, placebo-controlled trial to compare the effects of empagliflozin (a type of SLGT2 inhibitors) versus placebo (in a 1:1 ratio) in reducing hepatic fat content as measured by MRI-PDFF in NAFLD patients without DM. A total of 98 adult patients will be randomly sampled from the liver clinical in our local hospital. Empagliflozin 10mg daily will be given to the treatment arm. The placebo pill will be manufactured to be identical in appearance to the study drug. Eligible subjects will be followed up until week 52, and will undergo clinical, anthropometric and laboratory assessments (including liver function test and fasting blood) at baseline, week 6, 12, 26, 40 and 52. They will undergo LSM at baseline, week 26 and 52, and MRI-PDFF at baseline and week 52. The primary outcome will be a difference in change of liver fat content (measured by MRI-PDFF) at week 52 from baseline between the two groups. The secondary outcomes will be remission of steatosis (MRI-PDFF <5%) at week 52, reduction of liver fibrosis (LSM) at week 26 and 52, improvement of laboratory results (including liver transaminases and ductal enzymes, fasting glucose, HbA1c, lipid profile), improvement of anthropometric measurements, and combined cardiovascular and cerebrovascular events.

The study results will determine whether SGLT2 inhibitors can reduce hepatic steatosis and regress fibrosis in NAFLD patients without DM.

ELIGIBILITY:
Inclusion Criteria:

* Potential study subjects will first be screened by transient elastography for the presence of hepatic steatosis (defined as a measurement of controlled attenuation parameter [CAP] >= 248 db/M).
* They will be recruited into study if steatosis is >= 5% as confirmed by MRI-PDFF

Exclusion Criteria:

* DM (defined as hemoglobin A1c [HbA1c] >= 6.5% or fasting glucose >= 7.0 mmol/L)
* alcohol intake > 20g within past 2 years
* concurrent chronic liver diseases (including chronic viral hepatitis infection, autoimmune hepatitis, Wilson's disease, hemochromatosis, congestive hepatopathy, primary biliary cholangitis, primary sclerosing cholangitis, biliary tract obstruction)
* drug-induced liver disease
* usage of drugs that can lead to hepatic steatosis (e.g. steroids, amiodarone, valproate, methotrexate, tamoxifen)
* decompensated cirrhosis (including ascites, hepatic hydrothorax, variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, hepatopulmonary syndrome)
* history of malignancy including HCC
* recreational substance abuse
* pregnancy
* contraindications to empagliflozin use (estimated glomerular filtration rate [eGFR] <45mL/min/1.73m2 as measured by the MDRD equation, history of recurrent genitourinary tract infections, gangrene, or allergy)
* contraindications to MRI (e.g., claustrophobia, certain cardiac pacemakers, implanted medical devices with ferromagnetic properties).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content | week 52
  Difference in the change of liver fat content between the two groups at week 52 from the baseline as measured by MRI-PDFF

SECONDARY OUTCOMES:
Remission of steatosis | week 52
  Remission of steatosis (defined as MRI-PDFF < 5%) at week 52
Change of liver fat content | week 26 and 52
  Difference in the change of liver fat content between the two groups at week 26 and 52 from the baseline (CAP measured by transient elastography)
Changes of alanine aminotransferase (ALT) | week 52
  Changes of ALT at week 52
Changes of aspartate aminotransferase (AST) | week 52
  Changes of AST at week 52
Changes of alkaline phosphatase (ALP) | week 52
  Changes of ALP at week 52
Changes of gamma glutamyl transferase (GGT) | week 52
  Changes of GGT at week 52
Changes of fasting glucose | week 52
  Changes of fasting glucose at week 52
Changes of haemoglobin A1c (HbA1c) | week 52
  Changes of HbA1c at week 52
Changes of total cholesterol | week 52
  Changes of total cholesterol at week 52
Changes of low density lipoprotein (LDL) | week 52
  Changes of LDL at week 52
Changes of high density lipoprotein (HDL) | week 52
  Changes of HDL at week 52
Changes of body weight | week 52
  Changes of body weight at week 52
Changes of height | week 52
  Changes of height at week 52
Changes of body mass index (BMI) | week 52
  Changes of BMI at week 52
Changes of waist circumference | week 52
  Changes of waist circumference at week 52
Changes of systolic blood pressure | week 52
  Changes of systolic blood pressure at week 52
Changes of diastolic blood pressure | week 52
  Changes of diastolic blood pressure at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Ka Shing Cheung, MD, MPH, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong/Queen Mary Hospital, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No
IPD will be made available in the form of excel files upon request by other researchers

REFERENCES:
- [Derived] Cheung KS, Ng HY, Hui RWH, Lam LK, Mak LY, Ho YC, Tan JT, Chan EW, Seto WK, Yuen MF, Leung WK. Effects of empagliflozin on liver fat in patients with metabolic dysfunction-associated steatotic liver disease without diabetes mellitus: A randomized, double-blind, placebo-controlled trial. Hepatology. 2024 Oct 1;80(4):916-927. doi: 10.1097/HEP.0000000000000855. Epub 2024 Mar 27. PMID 38536017